CLINICAL TRIAL: NCT05882955
Title: Designing a Mixed-initiative Recipe Recommender App for Vegan and Vegetarian Sub-groups
Acronym: PERNUG
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: G-2021-4203-R5(AMD)
Record Dates: First submitted 2023-05-12; First posted 2023-05-31 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Mobile Applications
Keywords: app usage; recipe recommender acceptance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dietary app 1 (Experimental): Dietary app recommends high iron or iron focused recipes
  Interventions: Behavioral: Recipes consumption; Behavioral: Hydroponic unit
- Dietary app 2 (Sham Comparator): Dietary app recommends standard iron recipes
  Interventions: Behavioral: Recipes consumption; Behavioral: Hydroponic unit
- Hydroponic unit 1 (Experimental): Growing vitamin B12 biofortified plants in a hydroponic unit
  Interventions: Behavioral: Recipes consumption; Behavioral: Hydroponic unit
- Hydroponic unit 2 (No Intervention): No hydroponic unit given to participants

INTERVENTIONS:
Behavioral: Recipes consumption — Participants will eat one or two recipes a day for 17 weeks
  Arms: Dietary app 1; Dietary app 2; Hydroponic unit 1
Behavioral: Hydroponic unit — Participants will grow vitamin B12 biofortified plants for 17 weeks and consume (10 grams) of plant material for 11 weeks.
  Arms: Dietary app 1; Dietary app 2; Hydroponic unit 1

SUMMARY:
The goal of this study is to test the usability and applicability of a mobile application which recommends recipes. We will recruit up to 52 vegan/vegetarian participants in Belgium, and provide them with an iDOO hydroponic plant growing unit (https://www.idooworld.com/products/idoo-20pods-indoor-herb-garden-kit-hydroponics-growing-system-with-led-grow-light) as well as seeds and plant nutrients to grow certain herbs at home. Over a period of 17 weeks, participants will be asked to consume plants from the unit by following the recipes recommended by the app. The participants will then observe changes in their iron and vitamin B12 levels by following up with their GP and report the outcomes back to the researchers at three points during the study (week 0, week 6, and week 17). In addition, the participants will evaluate the usability of the app and the recipes recommended by the app.

DETAILED DESCRIPTION:
Iron is present in plant and animal-derived foods but the fractional absorption of iron from plant foods (that is the percent of iron absorbed from a consumed quantity) is often low (approx 10%) compared to iron from animal sources 25%-30%. It is therefore more challenging for vegans and vegetarians to achieve the Reference Nutrient Intake (RNI) for iron (8.7 mg/day for men over 18 and women over 50, 14.8 mg/day for women aged 18-50), and they are likely to absorb less of that iron and therefore are more likely to become iron depleted.

Plants do not synthesise vitamin B12 and unless fortified, plant-derived foods and beverages do not contain any vitamin B12. the RNI for vitamin B12 in the UK is 1.5 µg/day, therefore it is crucial that vegans and vegetarians take B12 supplements if they don't consume B12-fortified foods or find other ways of incorporating this vitamin into their diets.

Over a period of 17 weeks, participants will be asked to consume plants from the unit by following the recipes recommended by the app. The participants will then observe changes in their iron and vitamin B12 levels by following up with their GP and report the outcomes back to the researchers at three points during the study (week 0, week 6, and week 17). In addition, the participants will evaluate the usability of the app and the recipes recommended by the app.

ELIGIBILITY:
Inclusion Criteria

1. Healthy menstruating female with regular menstruation cycle over 18 years old.
2. Has been vegan, vegetarian or other diets that do not include the consumption of meat and fish for at least 1 year.
3. Willing to remain on a plant-based diet for the duration of the study.
4. Body Mass Index (BMI) between 18.5 - 40 kg/m2.
5. Lives in Belgium.
6. Willing to maintain a hydroponic unit at home and consume plants grown in the hydroponic unit (e.g., parsley, rocket, mizuna).
7. Access to a smartphone or online platform as well as access to the internet.

Exclusion Criteria

1. Those who have known allergies to the hydroponically grown salad greens (parsley, rocket, mizuna).
2. Pescatarian (consumes fish and seafood) and flexitarian (consumes meat intermittently) vegetarian.
3. Those with abnormal menstruation cycle time periods, <21 and >40-day
4. BMI < 18.5 kg/m2 (underweight) and > 40 kg/m2 (severely obese).
5. Those diagnosed or undergoing treatment for anaemia.
6. Currently pregnant or lactating.
7. Diagnosed medical conditions that may impact the study outcomes will be considered on an individual basis.
8. On a, or about to start, a diet programme such as the 5:2 programme (5:2 programme is where an individual would eat normally for five days a week, and fast for two days a week by reducing calorie consumption).
9. Unable to give written or verbal informed consent.
10. Participating in another dietary intervention study nor given blood in another dietary study in the last 3 months.
11. Any person related to or living with any member of the study team.
12. Those who are part of the Line Manager/supervisory structure of the Chief Investigator.
13. Those who have been asked to self-isolate or have been diagnosed with COVID-19 in the last 14 days. However, participants can be rescreened 7 days after the isolation period.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 52 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in serum ferritin after the dietary app intervention | Week: 0, 6/7 and 17
  Comparison of serum ferritin at baseline and after the intervention
Change of serum B12 after the hydroponic unit intervention | Week: 6/7 and 17
  Comparison of serum B12 at baseline and after the intervention

SECONDARY OUTCOMES:
App usability rating | Week: 6/7 and 17
  The usability of the mobile application will be scored on 100 using the System Usability Scale
Score on the Unified Theory of Acceptance and Use of Technology questionnaire | Week: 6/7 and 17
  The acceptance of the mobile application will be measured using the Unified Theory of Acceptance and Use of Technology questionnaire on a scale of 1 to 5.
Recipe recommendation performance | Week: 17
  The performance of the recipe recommendation system will be measured using the RESQUE questionnaire on a scale of 1 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Katrien Verbert, Principal Investigator — KU Leuven
Locations (1):
- Departement Computerwetenschappen, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No